CLINICAL TRIAL: NCT06790342
Title: Optimizing Treatment of Co-occurring Smoking and Unhealthy Alcohol Use Among PWH in Nairobi, Kenya
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB24-1626; 1R01CA288235-01A1 (NIH)
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: HIV; Tobacco Use; Alcohol Use Disorder
Keywords: HIV; Tobacco Cessation; Alcohol Reduction
MeSH Terms: conditions — Tobacco Use; Alcoholism; Tobacco Use Cessation | interventions — Cystine; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Cystine (CYT) + Positively Smoke Free (Experimental): Positively smoke free-- an 8 session tailored behavioral treatment for smoking cessation and alcohol reduction
  Cystine--used for smoking cessation and alcohol reduction
  Interventions: Drug: Cystine; Behavioral: Positively Smoke Free
- Experimental: Cystine + Standard of Care (Experimental): Cystine--used for smoking cessation and alcohol reduction
  Standard of Care--brief advice to quit provided in a standardized format bupropion--used for smoking cessation
  Interventions: Drug: Cystine; Other: Standard of Care
- Experimental: Placebo + Positively Smoke Free (Experimental): Positively smoke free-- an 8 session tailored behavioral treatment for smoking cessation and alcohol reduction
  Placebo--matched to bupropion
  Interventions: Behavioral: Positively Smoke Free; Other: Placebo
- Placebo Comparator: Placebo + Standard of Care. (Placebo Comparator): Placebo--matched to bupropion
  Standard of Care--brief advice to quit provided in a standardized format
  Interventions: Other: Placebo; Other: Standard of Care

INTERVENTIONS:
Drug: Cystine — Used for smoking cessation and alcohol reduction
  Arms: Experimental: Cystine (CYT) + Positively Smoke Free; Experimental: Cystine + Standard of Care
Behavioral: Positively Smoke Free — An 8 session tailored behavioral treatment for smoking cessation and alcohol reduction
  Arms: Experimental: Cystine (CYT) + Positively Smoke Free; Experimental: Placebo + Positively Smoke Free
Other: Placebo — Matched to cystine
  Arms: Experimental: Placebo + Positively Smoke Free; Placebo Comparator: Placebo + Standard of Care.
Other: Standard of Care — Standardized brief advice to quit smoking (standard of care)
  Arms: Experimental: Cystine + Standard of Care; Placebo Comparator: Placebo + Standard of Care.

SUMMARY:
People with HIV (PWH) smoke tobacco cigarettes and drink alcohol at higher rates than the general population, both in the US and internationally, including low- and middle-income countries. Now that effective antiretroviral therapy is available throughout most of the world, PWH are surviving long enough to manifest the lethal consequences of both their smoking and drinking. In this project, the investigational team aims to advance the knowledge and understanding of treatment strategies (i.e. individual intensive counseling ± pharmacotherapy with cytisine) that target both tobacco and alcohol use among PWH in Kenya, a resource constrained environment, and to generate outcome data that may benefit co-users of tobacco and alcohol throughout the world.

DETAILED DESCRIPTION:
This study was reviewed and approved for data analysis by the University of Chicago.

The research portion of this study was also submitted to and is pending approval from:

Board Name: AMREF ETHICAL AND SCIENTIFIC REVIEW COMMITTEE (ESRC) Board Affiliation: The AMREF ESRC is affiliated with AMREF Health Africa and accredited by National Commission for Science, Technology and Innovation (NACOSTI) since 200 Phone: +254 20 699 4000 Email: esrc.kenya@amref.org

Address:

Langata Road PO Box 27691-00506 Nairobi, Kenya

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed chart diagnosis of HIV
2. At least 18 years or age
3. Currently self-reports smoking (has smoked a cigarette within the past 7 days) and has expired air Carbon Monoxide (CO) 6ppm. Expired air CO provides an accurate indirect measure of carboxyhemoglobin (COHb) level and is a standard biochemical method for assessing a smoker's level of intake.
4. Motivation to quit smoking within the next 6 months (score 6-8 on the Abrams and Biener Readiness to Quit Ladder)
5. Meets criteria for heavy drinking: National Institute on Alcohol Abuse and Alcoholism (NIAAA) guidelines suggest gender-based criteria for heavy drinking but note that lower thresholds may be needed for people with a medical condition. PWH show increased physiologic injury and decreased survival at lower levels of alcohol consumption than those without HIV. Thus, we will use the lower limit for alcohol misuse/heavy drinking from the NIAAA guidelines for all study candidates, i.e. drinking 4+ drinks on a given day or >7 drinks/week over the past 30 days
6. Able to speak English (in Nairobi spoken English is near universal as English is an official language of Kenya)
7. Willingness to accept behavioral and/or pharmacologic tobacco and alcohol treatment
8. Willingness and ability to provide informed consent to participate.

Exclusion Criteria:

1. Current receipt of any tobacco or alcohol use behavioral or pharmacologic treatment
2. Previous allergic reaction or hypersensitivity to cytosine (CYT) (unlikely since CYT is not available in Kenya)
3. History of severe alcohol withdrawal symptoms in the past 12 months, including seizure or hallucinations
4. Pregnant, nursing, or becoming pregnant during the study
5. Current use of any medication that would interfere with the protocol in the opinion of the Medically Accountable Physician
6. Meets criteria for possible dementia by scoring below 10 on the Hopkins HIV Dementia Scale
7. Unstable psychiatric illness
8. Known plans to re-locate or travel away from the study site for more than two consecutive months during the study period
9. Expected survival of less than 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence abstinence (PPA) | 36 months
  Defined as self-reported no smoking in the past 7 days + Carbon Monoxide (CO)<7 ppm
Dried blood spot phosphatidylethanol (PEth) | 36 months
  PEth level of less than 50ng/dl for cessation from heavy drinking linked (P30D)
Timeline Follow-Back (TLFB) | 36 months
  denial of self-reported heavy drinking days (denying any prior 7-day period with >7 drinks or any single day with 4 drinks) for the past 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Seth Himelhoch, Principal Investigator — University of Chicago
Locations (2):
- Kenya (2):
  - Mathari National Teaching and Referral Hospital, Nairobi
  - Riruta Health Centre, Nairobi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rigotti NA, Benowitz NL, Prochaska J, Leischow S, Nides M, Blumenstein B, Clarke A, Cain D, Jacobs C. Cytisinicline for Smoking Cessation: A Randomized Clinical Trial. JAMA. 2023 Jul 11;330(2):152-160. doi: 10.1001/jama.2023.10042. PMID 37432430
- [Background] Himelhoch SS, Koech E, Omanya AA, Oduor P, Mchembere W, Masai TW, Bennett ME, Li L, Potts W, Ojoo S, Shuter J. Efficacy of Smoking Cessation Interventions among People with HIV in Kenya. NEJM Evid. 2024 Nov;3(11):EVIDoa2400090. doi: 10.1056/EVIDoa2400090. Epub 2024 Oct 22. PMID 39437141